CLINICAL TRIAL: NCT00581789
Title: Phase I Study of Erlotinib and Sunitinib in Non-small Cell Lung Cancer
Brief Title: Erlotinib and Sunitinib in NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pfizer (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2007-0063; CO05507; H-2007-0063 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2011-00549 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2012-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; sunitinib; erlotinib; phase 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Erlotinib 150mg PO daily + sunitinib 25mg PO daily (level 1) or 37.5mg PO daily (level 2)
  Interventions: Drug: erlotinib, sunitinib

INTERVENTIONS:
Drug: erlotinib, sunitinib — erlotinib 150mg PO daily + sunitinib 25mg PO daily (level 1) or 37.5mg PO daily (level 2)
  Other Names: Tarceva; OSI-774; Sutent; SU011248

SUMMARY:
* To determine the safety and maximally tolerated dose of sunitinib plus erlotinib in patients with non-small cell lung cancer (NSCLC).
* To determine response to sunitinib plus erlotinib in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven stage IIIB (with pleural effusion or pericardial effusion) or IV (either primary or recurrent) NSCLC (except squamous cell histology).
* Measurable disease per RECIST
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, hepatic and renal function
* ECOG performance status 0, 1 or 2.
* One and only one prior treatment with a chemotherapy regimen, including a platinum based regimen for advanced disease (Stage IIIB with malignant effusion or Stage IV).
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Female patients must be surgically sterile, postmenopausal or agree to use effective contraception during the period of therapy. Male patients must be surgically sterile or agree to use effective contraception during the period of therapy.

Exclusion Criteria:

* Squamous cell histology.
* History of untreated brain metastases
* Prior treatment with >1 systemic chemotherapy-based regimens for advanced disease (Stage IIIB with malignant effusion or Stage IV).
* Prior treatment with any receptor tyrosine kinase inhibitors, VEGF inhibitors, or other angiogenic inhibitors (including but not limited to bevacizumab, sunitinib, erlotinib, gefitinib, or thalidomide).
* Prior chemotherapy, radiation therapy, surgery, or investigational agent within 4 weeks prior to study entry, except palliative radiation therapy to a non-target lesions (must have been completed 2 weeks prior to study enrollment).
* Eligibility of patients receiving any medications or substances known to induce or inhibit CYP3A4 and /or with the potential to affect the activity or pharmacokinetics of sunitinib or erlotinib will be determined following review of their case by the Principal Investigator.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting therapy.
* Ongoing treatment with warfarin
* Prior treatment with high-dose chemotherapy requiring stem cell rescue.
* Prior irradiation to >25% of the bone marrow (whole pelvis = 25%).
* Diagnosis within prior 3 years of second malignancy, except basal cell carcinoma, squamous cell skin carcinoma or in situ carcinoma that has been completely treated without evidence of recurrent disease for 12 months.
* Current treatment on another therapeutic clinical trial or receipt of another investigative agent within 4 weeks of study entry.
* Any of the following within 12 months prior to starting study treatment: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus.
* Hypertension (>150/100mmHg) that cannot be controlled with standard antihypertensive agents.
* Ongoing cardiac dysrhythmias of grade >2, ≥ grade 3 atrial fibrillation, or QTc interval of >450 msec for males and >470 msec for females.
* Evidence of hemoptysis <4 weeks of starting study treatment.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality
* HIV-positive patients
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months

SECONDARY OUTCOMES:
Response rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu